CLINICAL TRIAL: NCT02658162
Title: A Randomized, Placebo-controlled, Prospective, Single-blind, Single Center Phase 2 Study of the Efficacy and Safety of SANGUINATE™ for Reduction of Delayed Graft Function in Recipients of a Donation After Brain Death Kidney Transplant
Brief Title: A Study on SANGUINATE™ for the Reduction of Delayed Graft Function in Kidney Transplant Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Prolong Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SGTP-003
Record Dates: First submitted 2016-01-12; First posted 2016-01-18 (Estimated); Last update posted 2018-05-25 (Actual); Status verified 2018-05

CONDITIONS: Delayed Function of Renal Transplant
MeSH Terms: interventions — PEGylated carboxyhemoglobin bovine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- SANGUINATE (Experimental): Two (2) infusions of SANGUINATE
  Interventions: Drug: SANGUINATE
- Normal Saline (Placebo Comparator): Two (2) infusions of Normal Saline
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: SANGUINATE — Two (2) infusions of 320 mg/kg of SANGUINATE at Baseline and Day 1
  Other Names: pegylated carboxyhemoglobin bovine
  Arms: SANGUINATE
Drug: Normal Saline — Two (2) infusions of Normal Saline at an equal volume to SANGUINATE at Baseline and Day 1.
  Arms: Normal Saline

SUMMARY:
Safety and efficacy study of SANGUINATE on reduction of delayed graft function (DGF) in patients who will be recipients of a donation after brain death (DBD) donor kidney.

DETAILED DESCRIPTION:
Sixty (60) adult subjects who will be recipients of a donation after brain death (DBD) donor kidney and who meet all eligibility criteria will be randomized 1:1 within 48 hours prior to transplant surgery to receive: two infusions of SANGUINATE at a dose of 320 mg/kg or placebo on the day of surgery and approximately 24 hours after surgery. Patients will be hospitalized for up to 5 days and the study duration will be 30 days.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and provide written informed consent.
2. Male or female subject at least 18 years of age.
3. Dialysis-dependent renal failure initiated at least 3 months prior to transplantation.
4. Subject is to be the recipient of a first kidney transplant from a deceased donor (brain death criteria).
5. Is able to receive intravenous infusions of study drug.
6. Anticipated donor organ cold ischemia time < 30 hours.
7. A calculated prediction of DGF risk of least 25%.
8. Females of childbearing potential must agree to use 2 forms of effective birth control regimen (at least one-barrier method) during the initial 30-day study period.
9. Male subjects must agree to use condoms or other suitable means of pregnancy prevention.

Exclusion Criteria:

1. Has received a blood transfusion of packed red blood cells (PRBC), other than with leukocyte-poor blood, within the 90-day period prior to screening.
2. Recipient of a live donor kidney or a kidney from a donation after cardiac death (DCD) donor.
3. Recipient of donor kidney preserved with normothermic machine perfusion.
4. Is scheduled to undergo multi-organ transplantation.
5. Has planned transplant of kidney(s) from a donor < 6 years of age.
6. Has planned transplant of kidneys that are implanted en bloc (dual kidney transplant).
7. Has planned transplant of dual kidneys (from the same donor) transplanted not en bloc.
8. Body Mass Index (BMI) > 38 kg/m2
9. Machine perfused preservation donor kidney.
10. Is scheduled for transplantation of a kidney from a donor who is known to have received an investigational therapy (under another Investigational New Drug) for ischemic/reperfusion injury immediately prior to organ recovery.
11. Is scheduled to receive an blood type-incompatible donor kidney.
12. Has undergone desensitization to remove antibodies prior to transplantation.
13. Total bilirubin > 1.5 mg per dL, transaminase more than twice the upper limit of normal or evidence of hepatic insufficiency
14. Has participated in an investigational study within the last 30 days or received an investigational product within 5 half-lives of the study drug administration, whichever is longest. Potential subjects participating in a strictly observational study or a study involving approved treatments should be discussed with the Medical Monitor.
15. Has a history of human immunodeficiency virus (HIV)
16. History or presence of active substance abuse (illicit drugs or alcohol) in the previous 6 months, as believed by the Investigator
17. Presence of ECG-based evidence of acute myocardial infarction, unstable angina, decompensated heart failure, third degree heart block or cardiac arrhythmia associated with hemodynamic instability
18. History or presence of any disease or psychiatric condition that in the Investigator's assessment that would increase the risk to subjects associated with study participation, drug administration or interpretation of results
19. History of biopsy-confirmed malignancy within 5 years of randomization, with the exception of adequately treated basal cell or squamous cell carcinoma in situ skin lesions, carcinoma of the cervix in situ, or early detected prostate cancer.
20. Female subject who is pregnant or breast feeding.
21. Has a positive T- or B-cell cross-match by NIH anti-globulin lymphocytotoxicity method, if performed.
22. Has a positive T- or B-cell cross-match AND donor specific anti-human leukocyte antigen (anti-HLA) antibody (DSA) detected by flow cytometry/Luminex based antigen-specific anti-HLA antibody testing, if performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02 (Estimated); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of delayed graft function (DGF) | 30 Days
  Reduction of delayed draft function will be measured by the number of dialysis sessions.
Participants With at Least One Occurrence of Safety Composite Endpoint by Treatment Group. | 30 Days
  Composite endpoint defined by changes in vital signs, electrocardiographic, biochemical, hematological, and urinalysis, graft loss, death and other reported adverse events and Graft Survival - 30 Days

SECONDARY OUTCOMES:
Proportion of subjects requiring dialysis for any reason in the first 7 days post-transplant | 7 Days
Proportion of subjects requiring dialysis only in the first 5 days post-transplant | 5 Days
Number of days of dialysis therapy. | 30 Days
Proportion of subjects with a fall in serum creatinine. | 7 Days
Proportion of subjects with a serum creatinine greater than 3 mg/dL, but who did not require dialysis by Day 5 post-transplant | 5 Days
Change in estimated creatinine clearance before and after kidney transplantation. | 30 Days
Change in estimated glomerular filtration rate before and after kidney transplantation. | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Hemant Misra, PhD, Study Director — Prolong Pharmaceuticals